CLINICAL TRIAL: NCT03672474
Title: Pilot Study Evaluating the Safety and Efficacy of a Photobiomodulation Prototype, REGEnLIFE RGn530 Device, on Cognitive Performances Evolution From Mild-to-moderate Alzheimer's Disease Patients
Brief Title: REGEnLIFE RGn530 - Feasibility Pilot
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid19 sanitary crisis
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECHMPL18_0075; 2018-A00404-51 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-08-03; First posted 2018-09-14 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Photobiomodulation; Innovative Therapy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photobiomodulation REGEnLIFE RGn530 device group (Experimental)
  Interventions: Device: Photobiomodulation REGEnLIFE RGn530 device
- Sham REGEnLIFE RGn530 device group (Sham Comparator)
  Interventions: Device: SHAM REGEnLIFE RGn530 device

INTERVENTIONS:
Device: Photobiomodulation REGEnLIFE RGn530 device — For the photobiomodulation group the device is set up and activated. REGEnLIFE RGn530 medical device will follow EC labelling if proven to be safe and effective
  Arms: Photobiomodulation REGEnLIFE RGn530 device group
Device: SHAM REGEnLIFE RGn530 device — For the photobiomodulation group the device is set up and not activated. REGEnLIFE RGn530 medical device will follow EC labelling if proven to be safe and effective
  Arms: Sham REGEnLIFE RGn530 device group

SUMMARY:
REGEnLIFE RGn530 is a photobiomodulation medical device, consisting in a modular helmet and abdominal panel, composed of near-infrared low-level lasers (LLLT), near-infrared and red LEDs as well as a static magnetic field. RGn device application on both head and abdomen have demonstrated striking efficacy in preclinical studies. The investigator's results clearly indicated that RGn treatment produces a normalization of all parameters that are strongly modified in the model, including memory performances associated to oxidative stress, neuroinflammation or apoptosis markers, microbiota composition and specific markers related to the amyloid or tau processes (Blivet et al., Alzheimers Dement (NY), 2018).

Following such promising results, this pilot clinical study will evaluate the safety and efficacy of REGEnLIFE RGn530 device on cognitive performances evolution from mild-to-moderate Alzheimer's disease patients. The double-blind, randomized, monocentric sham-controlled clinical trial will be performed at the CHU de Montpellier. 64 patients will be enrolled: 32 in photobiomodulation group and 32 in sham group. Each patient will follow 8 weeks of treatment with 5 sessions of 25min per week (total of 40 sessions) and will undergo, for a total period of three months, series of clinical examinations including cognitive evaluation, biological and electrophysiological analyses, sleep recordings, and imaging assessments.

REGEnLIFE RGn530 medical device will follow EC labelling if proven to be safe and effective. In the light of anti-amyloid therapeutic approaches lack of success, RGn530 dual treatment is hoped to be particularly valuable as an innovative and extensive treatment strategy for AD.

DETAILED DESCRIPTION:
Design : Prospective monocentric double-blind pilot study with 2 parallel groups of 32 patients. One with photobiomodulation (device set up and activated), the other with placebo-sham procedure (device set up but not activated). The study will consist of an inclusion visit (V0, D-30 to D-10), a photobiomodulation start visit (V1, D0), followed by 3 follow-up visits (V2 to D30, V3 to D60 and V4 to D90).

Dispositive : Photobiomodulation device developed by REGEnLIFE, RGn530 consisting of a modular helmet and an abdominal modular panel each comprising modules composed of low intensity infrared lasers (LLLT - Low Level Laser Therapy), infrared and red LEDs and a static magnetic field. The helmet and abdominal panel devices are connected to a steering console. Activation of the device will be done by personnel trained for this purpose by REGEnLIFE.

Originality and innovation : This study proposes to evaluate a new medical photobiomodulation device in the field of neurodegenerative diseases. These techniques have shown positive and promising results in the following areas: wound healing, pain management, inflammation, tissue regeneration, and the following disciplines: neuropsychiatry, dermatology and neurology.

Photobiomodulation is a technology of the same family as phototherapy, also called LLLT (Low Level Laser Therapy). It can be defined as the directional use of monochromatic or polychromatic light from low energy lasers and / or LEDs, in wavelengths included in the visible, infrared and near infrared, to modulate a function or induce a therapeutic effect in an athermal, non-invasive and non-destructive manner.

This pilot study aims to evaluate the efficacy and safety of this new non-invasive pre-marking device in patients with mild to moderate AD. To date, no study has been published with this device on this typology of patients.

Duration of treatment : 8 weeks with 5 sessions of 25 minutes per week, for a total of 40 sessions.

Study population : Patients with international AD diagnosis criteria according to McKhann et al., 2011 at mild to moderate stage (MMSE score between 16-26), having agreed and signed free and informed consent to participate in this study, without contraindications to the carrying out of the complementary investigations necessary for the evaluation of the efficiency and the tolerance of the RGn530.

Schedule of visits : Each patient will be followed for 3 months at the rate of 5 visits: inclusion V0 (D-10 to D-30), V1 (D0), V2 (M1), V3 (M2) and V4 (M3).

Number of patients : 64 patients will be included in this study: 32 in the photobiomodulation group and 32 in the placebo-sham group.

Duration of patient follow-up : Each patient will be followed for a total duration of 3 months with visits involving clinical, biological, electrophysiological, imaging, tests and questionnaires to assess the efficacy and tolerance of RGn530.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or Female ;
* Age between 55-85 years old ;
* Diagnostic of AD according to international criteria of McKhann et al., 2011 [1] ;
* Mild-to-moderate Alzheimer's disease stage with MMSE score between 16 and 26 ;
* Symptomatic treatments specific to AD (Memantine, acetylcholinesterase inhibitors) and pyshotropic treatments (anxiolytics, anti-depressants, neuroleptics) are allowed but must be maintained at fixed doses during the 4 weeks previous to inclusion and during all the study length ;
* Patient approval for biological, eletrophysiological and imaging tests ;
* Enough availability to participate daily to the proposed treatment sessions ;
* Given informed, free consent, written and signed by participant and investigator (at the latest on the day of inclusion and before any examination needed for the research) ;
* Affiliated to social security regime or beneficiary of such a regime ;
* Patient given approval to perform a second lumbar puncture (without contraindication) if tests results and/or neurological follow-up need a CSF test for biomarkers ;

Exclusion Criteria:

* Exclusion criteria:
* Clinical and paraclinical details insufficient for AD diagnostic ;
* Genetic form of AD (genetic mutation characterized) ;
* No caregiver to complete neuropsychological scales and evaluation forms ;
* Patient living in a medical institution ;
* Illiteracy or inability to perform psycho-behavioral tests ;
* Physical or neurosensory problems susceptible to interfere with tests
* Contraindication or refusal to perform MRI imagerie examinations, PET-FDG, P300 and/or actimetry tests ;
* Patient carrying a pacemaker device or a ferromagnetic compound ;
* Short-term life-threatening pathologies (evolutive cancer, unstable cardiac failure, liver or kidney failure, severe respiratory insufficiency) ;
* Chronic psychosis or psychotic episodes ;
* Alcohol or drug addiction ;
* Epilpesy or other non-neurodegenerative diseases of the central nervous system ;
* Deficits in B12 and non-supplemented folic acid levels ;
* Untreated hypothyroidism ;
* Major skin lesions on treatment application regions (possibility to apply a bandage during the treatment if minor lesions) ;
* Recent major chirurgical intervention at the abdomen in the past three month before inclusion ;

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Orientation (time and space) score (10 items) from the Mini Mental Scale Examination (MMSE) | Month 2
  Mini Mental State Examination (MMSE) is a global cognition assessment (score between 0-30) Folstein MF, Folstein SE, McHugh PR. "Mini Mental State" a practical method for grading the cognitive state of patients for the clinicians. J Psychiat Res. 1975;12:189-19.
Sum of free recall (sum of the three learning tests) and of cued recall (sum of free recall and indexed recall) from the Free and Cued Selective Reminding Test (FCSRT) | Month 2
  Free Cued Selective Remainding Test (FCRST) is a memory test
  1. Grober E, Sanders AE, Hall C, Lipton RB. Free and cued selective reminding identifies very mild dementia in primary care. Alzheimer Dis Assoc Disord. 2010;24:284-90. ; 2. Mélissa Dion, Olivier Potvin, Sylvie Belleville, Guylaine Ferland, Mélanie Renaud, Louis Bherer, Sven Joubert, Guillaume T. Vallet, Martine Simard, Isabelle Rouleau, Sarah Lecomte, Joël Macoir & Carol Hudon (2014): Normative Data for the Rappel libre/Rappel indicé à 16 items (16-item Free and Cued Recall) in the Elderly Quebec-French Population, The Clinical Neuropsychologist ; 3. Van der Linden et al. L'épreuve de rappel libre / rappel indicé à 16 items (RL/RI-16), 2004
(3) Digit symbol Substitution test (WAIS-IV coding test) | Month 2
  Digit symbol Substitution test (WAIS-IV coding test) is an executive function assessment (score between 0-135)
  1.Wechsler, D., Kaplan, E., Fein, D., Kramer, J., Morris, R., Delis, D., & Maelender, A. (2003). Wechsler intelligence scale for children: Fourth edition (WISC-IV) [Assessment instrument]. San Antonio, TX; Pearson
(4) 2-minutes Category naming test | Month 2
  Category naming test (CNT) is a language test
  1.Cardebat D, Doyon B, Puel M, Goulet P, Joanette Y. Formal and semantic lexical evocation in normal subjects. Performance and dynamics of production as a function of sex, age and educational level. Acta Neurol Belg 1990

SECONDARY OUTCOMES:
MATTIS | Month 3
  MATTIS Dementia Rating Scale (MDRS) is a global cognitive assessment (score between 0-144)
  1. Schmidt R, Freidl W, Fazekas F, Reinhart B, Grieshofer P, Koch M, et al. The Mattis Dementia Rating Scale. Normative data from 1,001 healthy volunteers. Neurology. 1994;44:964-6. ; 2. Monica Lavoie , Brandy Callahan , Sylvie Belleville , Martine Simard , Nathalie Bier , Lise Gagnon , Jean-François Gagnon , Sophie Blanchet , Olivier Potvin , Carol Hudon & Joël Macoir (2013) Normative Data for the Dementia Rating Scale-2 in the French-Quebec Population, The Clinical Neuropsychologist, 27:7, 1150-1166
Trail Making Test A and B | Month 3
  Cognitive Assessment
ADAS-Cog | Month 3
  Alzheimer Disease Assessment Scale-Cognition (ADAS-Cog) is a global cognitive assessment (score between 0-70)
  1. Doraiswamy PM, Krishen A, Stallone F, Martin WL, Potts NL, Metz A, et al. Cognitive performance on the Alzheimer's Disease Assessment Scale: effect of education. Neurology. 1995;45:1980-4. ; 2. 1.Mohs et al. Development of Cognitive Instruments fort Use in Clinical Trials of Antidementia Drgus : Adiitions to the Alzheimer's Disease Assessment Scale That Broaden Its Scope, 1997
Clinical Dementia Rating | Month 3
  Clinical Dementia Rating (CDR) score, Questionnaire assessing general well-being, cognitive function (score between 0-5)
  1. Morris, J. C. (1997). Clinical dementia rating: a reliable and valid diagnostic and staging measure for dementia of the Alzheimer type. International psychogeriatrics, 9(S1), 173-176. ; 2. HUGONOT-DIENER L. La consultation de gériatrie. Masson. 2001
IADL 8 items | Month 3
  Instrumental Activities Of Daily Living (IADL) scale, Questionnaire assessing general autonomy (between 0-8) Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969;9:179-86.
Biological Parameters in blood | Month 2
  Level of blood plasma marker Hemoglobin (g/dL)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Erythrocytes (1012/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Platelets (109/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Leukocytes (109/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Neutrophilic Polynuclear (109/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Polynuclear Eosinophils (109/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Polynuclear Basophils (109/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Lymphocytes (109/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Monocytes (109/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Glycemia (blood glucose) (mmol/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Total Cholesterol (mmol/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker HDL Cholesterol (mmol/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker LDL Cholesterol (mmol/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Triglycérides (g/L)
Biological Parameters in blood | Month 2
  Level of marker Serum Glutamate Pyruvate Transaminase (SGPT) (UI/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Creatinine (µmol/ L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker C reactive protein (mg/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Thyroid Stimulating Hormon (TSH) (µUI/mL)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Cobalamin (B12 Vitamin) (ng/L)
Biological Parameters in blood | Month 2
  Level of blood plasma marker Folates (µg/L)
Biological Parameters in CSF | Month 2
  Level of CSF marker protein Aβ42 (pg/ml) Level of CSF marker protein Aβ40 (pg/ml) Level of CSF marker protein Tau (pg/ml) Level of CSF marker protein P-tau (pg/ml)
Electrophysiological Parameter | Month 2
  Wave P300, cerebral activity at 300ms after a stimulus. Analysis of the Amplitude (µV) of the Event-Related Potential (ERP) according to standardized protocol
Electrophysiological Parameter | Month 2
  Wave P300, cerebral activity at 300ms after a stimulus. Analysis of the Latency (ms) of the Event-Related Potential (ERP) according to standardized protocol
Electrophysiological Parameter | Month 2
  Wave P300, cerebral activity at 300ms after a stimulus. Analysis of the antero-posterior gradient (µV) of the Event-Related Potential (ERP) according to standardized protocol
Actimetry Activity Parameter | Month 2
  Activity parameter measuring by alternating plot daytime activity / nocturnal rest, througt an Actimetry Device. The patient will wear actigraphy bracelet during 10 days that will enable to record its movements. The report based on the recording will provide an assessment of night sleep duration.
Actimetry Activity Parameter | Month 2
  Activity parameter measuring by alternating plot daytime activity / nocturnal rest, througt an Actimetry Device. The patient will wear actigraphy bracelet during 10 days that will enable to record its movements. The report based on the recording will provide an assessment of sleep efficiency.
Actimetry Activity Parameter | Month 2
  Activity parameter measuring by alternating plot daytime activity / nocturnal rest, througt an Actimetry Device. The patient will wear actigraphy bracelet during 10 days that will enable to record its movements. The report based on the recording will provide an assessment of daytime somnolence
Morphological MRI 1.5T hippocampal Scheltens volumetry | Month 2
  Imaging
Imaging Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) values in regions of interest | Change from baseline at 3 months
  To determine if after the treatment, patients with Alzheimer's disease will have changes in regions of interest

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Gui de Chauliac, Montpellier, France

IPD SHARING:
Plan to Share IPD: No